CLINICAL TRIAL: NCT06524206
Title: An Awareness, Courage, and Love Intervention to Help Chinese Older Adults in the Post-pandemic Era: A Pilot Randomised Controlled Trial
Brief Title: An Awareness, Courage, and Love Intervention to Help Chinese Older Adults in the Post-pandemic Era
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caritas Institute of Higher Education (Other)
Responsible Party: Principal Investigator, Stephen Cheong Yu Chan, Assistant Professor, Caritas Institute of Higher Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CIHE
Record Dates: First submitted 2024-07-22; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Loneliness; Depression; Anxiety; Social Connectedness; Subjective Well-being; Psychological Intervention; Older Adults
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awareness, Courage, and Love intervention (Experimental): The Awareness, Courage and Love intervention will consist of a single 120-minute online session delivered in a group format via a videoconferencing application (e.g., Zoom). The theme of the session will evolve around "making friends and being seen" to reinforce the appetitive functions of social connection.
  Interventions: Behavioral: The Awareness, Courage and Love Intervention
- Waitlist control group (No Intervention): Waitlist control group will not receive the intervention

INTERVENTIONS:
Behavioral: The Awareness, Courage and Love Intervention — Derived from Functional Analytic Psychotherapy (FAP), the Awareness, Courage, and Love (ACL) Intervention brings the FAP principles to a broader population. In the ACL model, awareness is defined as engaging in mindful awareness of one's self (feelings, needs, values), other individuals, and the context in which interactions are taking place. Courage is defined as engaging in authentic, vulnerable self-disclosures (e.g. struggles, appreciation), and asking for what one wants and needs. Love is defined as providing empathically accurate responsiveness, including provision of safety, validation, and giving the other person what they have asked for when possible.
  Arms: Awareness, Courage, and Love intervention

SUMMARY:
The purpose of this study is to explore the potential effectiveness of a one-session online Awareness, Courage, and Love intervention for reducing loneliness, depression and anxiety symptoms, and enhancing social connectedness and subjective well-being among older adults. the study also aims to estimate the effect sizes of the Awareness, Courage, and Love intervention.

DETAILED DESCRIPTION:
The recruitment process will commence with referrals from local community organizations. Eligible individuals will be provided with detailed information about the study, and informed consent will be obtained from those willing to participate. After the confirmation of participant recruitment, a randomization process will be implemented to ensure the equitable distribution of participants between the intervention and waitlist control groups. An independent researcher will generate computer-generated random codes for group assignment, and these codes will be securely sealed in opaque envelopes. The envelopes will be sequentially numbered, and the randomization process will remain blinded throughout to prevent bias. Participants will be notified via email or text for the details of the condition they are assigned, and their willingness to engage in both the intervention and data collection will be confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. aged 60 years or older and dwelling in the community;
2. able to communicate in Cantonese;
3. have access to the internet and videoconferencing devices such as a mobile phone;
4. able to give informed consent to participate.

Exclusion Criteria:

1. severe emotional distress based on PHQ-4 screening assessment or presenting an imminent suicidal risk;
2. known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia/significant cognitive impairment;
3. illiterate;
4. difficulty in communication.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline on the Inclusion of Others in Self (IOS) at Immediately post-intervention and One-month post-intervention follow-up | Baseline, Immediately post-intervention and One-month post-intervention follow-up
  The single-item Inclusion of Others in the Self (IOS) scale is to measure how close the respondent feels with another person or group. Respondents choose a pair of photos from seven with different degrees of overlap. Possible scores range from 1 (No overlap) to 7 (Most overlap).

SECONDARY OUTCOMES:
Changes from Baseline on the 6-item de Jong Gierveld loneliness scale at Immediately post-intervention and One-month post-intervention follow-up | Baseline, Immediately post-intervention and One-month post-intervention follow-up
  The 6-item De Jong Gierveld Loneliness Scale is a reliable and valid measurement instrument for overall, emotional, and social loneliness. The possible range of scores is from 0 (Least lonely) to 6 (Most lonely).
Changes from Baseline on the Patient Health Questionnaire (PHQ-9) at Immediately post-intervention and One-month post-intervention follow-up | Baseline, Immediately post-intervention and One-month post-intervention follow-up
  The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression over the last 2 weeks. The interpretation of total scores ranges from 1-4 (Minimal depression) to 20-27 (Severe depression).
Changes from Baseline on the Generalized Anxiety Disorder 2-item (GAD-2) at Immediately post-intervention and One-month post-intervention follow-up | Baseline, Immediately post-intervention and One-month post-intervention follow-up
  The GAD-2 is a very brief and easy to perform initial screening tool for generalized anxiety disorder over the last 2 weeks. The possible scores range from 0 to 6. Higher scores are associated with higher levels of anxiety. A score of 3 points or more suggests possible anxiety.
Changes from Baseline on The World Health Organisation- Five Well-Being Index (WHO-5) at Immediately post-intervention and One-month post-intervention follow-up | Baseline, Immediately post-intervention and One-month post-intervention follow-up
  The WHO-5 is a short self-reported measure of current mental wellbeing. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Cheong Yu Chan, Dr, Principal Investigator — Caritas Institute of Higher Education
Locations (1):
- Caritas Institute of Higher Education, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No